CLINICAL TRIAL: NCT00434889
Title: Factors Associated With Falls and Near-Falls in Community Dwelling Older Adults With Early-Stage Dementia
Brief Title: A Study of Why People With Early Memory Problems Fall or Almost Fall
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Vanina Dal Bello-Haas, PhD, PT, Associate Professor, School of Physical Therapy, University of Saskatchewan
Other Study IDs: BIO-REB 06-181
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Dementia; Falls; Near-Falls
Keywords: dementia; falls; risk factors
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Memory problems
- 2: No memory problems

SUMMARY:
The purpose of this study is to identify the factors that are associated with falls and near falls in community-dwelling older adults with early-stage dementia.

DETAILED DESCRIPTION:
The specific objectives of this six month study are to: characterize falls and near-falls in community dwelling older adults with early-stage dementia; determine which potentially modifiable physical fall risk factors contribute to falls and near-falls in older adults with early-stage dementia; examine the relationship between dementia sub-type, medical and neuropsychological factors, balance and gait, and falls and near-falls in community dwelling older adults with early-stage dementia.

ELIGIBILITY:
Inclusion Criteria:

* males or females over the age of 50 with early-stage dementia as described by Global Deterioration Scale levels 2,3,4 or 5.

Exclusion Criteria:

* subjects who have a medical condition that significantly predispose them to falls (Meneire's disease or Parkinson's disease)
* subjects without a caregiver/spouse to assist with the completion of a Fall Diary
* subjects unable to stand independently or safely walk a short distance either unaided or with the support of an assistive device
* subjects unable to safely complete the balance and gait evaluations.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-08; Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vanina Dal Bello-Haas, Ph.D, Principal Investigator — University of Saskatchewan
Locations (1):
- School of Physical Therapy, University of Saskatchewan, Saskatoon, Saskatchewan, Canada